CLINICAL TRIAL: NCT02116036
Title: Rivaroxaban in Antiphospholipid Syndrome Pilot Study: A Multicenter Feasibility Study of Rivaroxaban for Patients With Antiphospholipid Syndrome and Prior Arterial or Venous Thrombosis
Brief Title: Rivaroxaban for Antiphospholipid Antibody Syndrome
Acronym: RAPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Bayer (Industry); Hamilton Health Sciences Corporation (Other); Jewish General Hospital (Other); University of Alberta (Other); The Ottawa Hospital (Other); Queen Elizabeth II Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: G-13-0002011
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Antiphospholipid Antibody Syndrome
Keywords: Antiphospholipid Antibody Syndrome; Rivaroxaban; Thromboembolism; Bleeding; Feasibility
MeSH Terms: conditions — Antiphospholipid Syndrome; Thromboembolism; Hemorrhage | interventions — Rivaroxaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rivaroxaban (Experimental): Rivaroxaban 20mg po daily
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: Rivaroxaban
  Other Names: Xarelto

SUMMARY:
The antiphospholipid antibody syndrome (APS) is a syndrome associated with excessive blood clotting (thrombosis). APS is among the most common cause of heart attack and stroke in patients under the age of 50 and is particularly prevalent in patients with autoimmune conditions. Patients with APS and prior thrombosis require lifelong anticoagulant therapy to prevent recurrent clots; such therapy is currently provided with warfarin. Warfarin requires frequent bloodwork monitoring, and many medications or foods can alter its effect, which can put people either at increased risk for clotting or bleeding. Rivaroxaban is a new mediation that prevents blood clots that does not require bloodwork monitoring and that has fewer interactions. This study is a pilot feasibility study which will: 1) examine our ability to identify 150 eligible APS patients; 2) measure our ability to obtain consent from 135 of these patients; and 3) test our hypothesis that we can obtain 95% compliance with daily rivaroxaban administration. The investigators propose to treat eligible patients with rivaroxaban 20 mg once daily. Patients will be followed for a minimum of one year and their rates of bleeding and thrombosis will be monitored as secondary outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Prior objectively-confirmed venous thrombosis, irrespective of history of arterial thrombosis
* Two or more prior positive APS serological evaluations at least 12 weeks apart
* Current treatment with warfarin administered to achieve an INR of 2.0 to 3.0, rivaroxaban or dabigatran at any dose currently used for secondary prophylaxis of thrombosis, or short term therapeutic dose LMWH (for example, for the treatment of recently diagnosed deep vein thrombosis). Patients not currently receiving anticoagulation but in whom anticoagulation is mandated, may also be enrolled if a 20 mg rivaroxaban dose would be appropriate

Exclusion Criteria:

* Prior recurrent thrombosis while taking warfarin with a demonstrated INR of 2.0 to 3.0, or prior recurrent thrombosis while receiving dabigatran or rivaroxaban
* History of isolated arterial thrombosis (no history of venous thrombosis) pending CTA approval by Health Canada
* Need for continued treatment with both aspirin (irrespective of dose) AND clopidogrel
* Pregnancy or planned pregnancy during the study period; women who may become pregnant will be required to utilize reliable contraceptive measures while on study drug
* Chronic kidney disease with calculated GFR < 30mL/min
* Geographic inaccessibility
* Age < 18 years
* Inability or failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2014-09; Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of identification for enrolment | 18 months
  The investigators define success as the ability to identify 150 eligible patients at 6 clinical centres over 18 months.
Feasibility of Consent | 18 months
  The investigators define success as a consent rate of 90% (thus, if we identify 150 patients, at least 135 will provide consent).
Compliance | Minimum of one year for all subjects
  The investigators define success as a patient missing fewer than 5% of days with pill administrations, as measured by pill counts.

SECONDARY OUTCOMES:
Bleeding | Minimum of one year for all subjects
  The investigators will collect and report the rates of minor bleeding (clinically apparent bleeding that does not meet the criteria for major), and major and fatal bleeding. Major bleeding will be defined by International Society of Thrombosis and Hemostasis criteria.
Thrombosis | Minimum of one year for all subjects
  The investigators will collect and report the rates of objectively-confirmed venous and arterial thrombosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly J Legault, MD, Principal Investigator — St. Joseph's Healthcare Hamilton, Hamilton Health Sciences; Mark A Crowther, MD, MSc, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (6):
- Canada (6):
  - University of Alberta Hospital, Edmonton, Alberta
  - Queen Elizabeth II Hospital, Halifax, Nova Scotia
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Jewish General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Legault K, Blostein M, Carrier M, Khan S, Schulman S, Shivakumar S, Wu C, Crowther MA. A single-arm feasibility cohort study of rivaroxaban in antiphospholipid syndrome. Pilot Feasibility Stud. 2020 Apr 25;6:52. doi: 10.1186/s40814-020-00594-1. eCollection 2020. PMID 32346486